CLINICAL TRIAL: NCT05770505
Title: Effect E-health Based Exercise Intervention After COVID-19
Brief Title: Use of E-health Based Exercise Intervention After COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 479316
Record Dates: First submitted 2023-03-13; First posted 2023-03-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise (Experimental)
  Interventions: Behavioral: Exercise training using an e-health tool
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Exercise training using an e-health tool — Experimental: Exercise training will be guided by using the e-health tool MIA Health, with the possibility for digital communication between the participants and study personnel The participants will receive wearables that record heart rate. Participants will be encouraged to achieve 100 Activity Quotient (AQ) equivalents per week Control: No follow-up
  Arms: Supervised exercise

SUMMARY:
Reduced subjective and objective functional capacity performance are reported after COVID-19 in a large proportion of subjects. The aim of this study is to examine the feasibility and effect of using an e-health tool for guidance and tracking of exercise training in a general population of adults previously infected by COVID-19.

DETAILED DESCRIPTION:
Both hospitalized and non-hospitalized persons who have undergone extensive multi-disciplinary rehabilitation programs report significantly improved physical function after rehabilitation. Exercise training may be the key intervention to improve fitness and subjective complaints such as fatigue, low physical fitness and dyspnea after COVID-19 infection. However, traditional group-based exercise training or self-training programs at fitness centers have been shut down during the pandemic, and home-based interventions are warranted. To overcome the limitations and costs of a fitness center/personal trainer-based intervention study, more knowledge on the effectiveness and efficacy of using an e-Health system to recruit, train and monitor participants after illness are needed.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have undergone COVID-19 disease
* People who struggle to be physically active enough as a result of corona disease
* People who experience reduced physical fitness as a result of corona disease

Exclusion Criteria:

-- more than 100 AQ per week (calculated from self-reported activity level)

* uncontrolled hypertension (high blood pressure) (over 200/110).
* symptomatic valve failure, hypertrophic cardiomyopathy, unstable angina, pulmonary
* hypertension, heart failure and/or severe rhythm disturbances
* cancer that makes participation impossible or exercise contraindicated. Considered individually in consultation with the attending physician.
* chronic contagious infectious diseases.
* Participates in other studies that are not compatible with participation in this project
* Post-exertional symptom exacerbation (PESE)/post-exertional malaise (PEM)/post-exertional neuroimmune exhaustion (PENE).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | After 6 months intervention
  Peak oxygen uptake
Feasibilty | After 6 months intervention
  Measured as acceptability and adherence

SECONDARY OUTCOMES:
Lung function | After 6 months intervention
  Spirometry
Quality of life | After 6 months intervention
  Questionnaires (RAND-12)

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Stensvold Stensvold, Principal Investigator — Dorthe Stensvold, Professor, NTNU
Locations (1):
- Norwegian University of Science and Technology, Faculty of medicine, Department of circulation and medical imaging,, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided